CLINICAL TRIAL: NCT06820554
Title: Thyroid Dysfunction Induced by Radiotherapy Treatment in Patients with Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, fatmaelzahraa mohamed said, residant doctor, Assiut University
Other Study IDs: TD radio brest cancer
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Brest Cancer
Keywords: Thyroid dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- brest cancer: breast cancer patients who will be indicated for postoperative ( mastectomy /BCT) adjuvant radiotherapy who are>18 yrs old breast cancer ( pathological proved ) Stage II/III breast cancer High risk local recurrence ( LVI/ G3/ LN positive) Non metastatic breast cancer

SUMMARY:
Breast cancer is the most common cancer and second most common cause of cancer death among US women,. External beam radiation therapy (RT) that involves the breast and regional lymph nodes, including axillary and supraclavicular (SCV) lymph nodes, has been demonstrated to decrease the risk of local recurrence and improve long-term survival in high-risk breast cancer patients .

However, RT-induced toxicities to adjacent normal tissues can lead to serious morbidity in cancer survivors .

The thyroid regulates the body's metabolism via producing thyroxine (T4) and triiodothyronine (T3) hormones. As the thyroid is sensitive to RT, radiation-induced thyroid disorders have been reported in cancer patients who received radiation in the cervical or SCV regions .

In breast cancer patients, RT to the SCV area has been associated with a higher incidence of Hypothyriodism, particularly in younger patients This complication may be associated with radiation-induced thyroid volume reduction .

Recent studies,have reported a significant decrease in thyroid volume (14-30 %) in patients with laryngeal or nasopharyngeal carcinoma (NPC), suggesting an association between HT and post-RT thyroid atrophy .

Little is known about the changes of thyroid gland volume based on local thyroid gland radiation dose and its correlations with incidence of HT.

Our study aim the changes in thyroid volume of breast cancer patients who received RT to the SCV nodal area, to evaluate RT-induced thyroid gland evolution based on local radiation dose. We then assessed the association between thyroid volume changes and the incidence of post-RT Hypothyrodism in breast cancer patients.

the aim of the study to diagnose subclinical hypothyroidism and biochemical changes in thyroid function after radiotherapy for breast cancer

DETAILED DESCRIPTION:
Breast cancer is the most common cancer and second most common cause of cancer death among US women,. External beam radiation therapy (RT) that involves the breast and regional lymph nodes, including axillary and supraclavicular (SCV) lymph nodes, has been demonstrated to decrease the risk of local recurrence and improve long-term survival in high-risk breast cancer patients .

However, RT-induced toxicities to adjacent normal tissues can lead to serious morbidity in cancer survivors .

The thyroid regulates the body's metabolism via producing thyroxine (T4) and triiodothyronine (T3) hormones. As the thyroid is sensitive to RT, radiation-induced thyroid disorders have been reported in cancer patients who received radiation in the cervical or SCV regions .

In breast cancer patients, RT to the SCV area has been associated with a higher incidence of Hypothyriodism, particularly in younger patients This complication may be associated with radiation-induced thyroid volume reduction .

Recent studies,have reported a significant decrease in thyroid volume (14-30 %) in patients with laryngeal or nasopharyngeal carcinoma (NPC), suggesting an association between HT and post-RT thyroid atrophy .

Little is known about the changes of thyroid gland volume based on local thyroid gland radiation dose and its correlations with incidence of HT.

Our study aim the changes in thyroid volume of breast cancer patients who received RT to the SCV nodal area, to evaluate RT-induced thyroid gland evolution based on local radiation dose. We then assessed the association between thyroid volume changes and the incidence of post-RT Hypothyrodism in breast cancer patients.

the aim of the study to diagnose subclinical hypothyroidism and biochemical changes in thyroid function after radiotherapy for breast cancer

ELIGIBILITY:
Inclusion Criteria:

* >18 yrs old breast cancer ( pathological proved )
* Stage II/III breast cancer
* High risk local recurrence ( LVI/ G3/ LN positive)
* Non metastatic breast cancer

Exclusion Criteria:

* Thyriod dysfunction of any othe cause( no known pretreatment primary thyroid disease or dysfunction; no prior thyroid surgery; and no prior RT that involved the hypothalamic-pituitary axis or thyroid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breast cancer patients who will be indicated for postoperative ( mastectomy /BCT) adjuvant radiotherapy
Sampling Method: Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
incidence of subclinical hypothyroidism | 3 months
  subclinical hypothyroidism after radiotherapy for breast cancer